CLINICAL TRIAL: NCT03832400
Title: A Phase 1b, Placebo-controlled, Study of the Safety and Efficacy of MET-2 in Patients With Ulcerative Colitis
Brief Title: Safety and Efficacy of Microbial Ecosystem Therapeutic-2 (MET-2) in Patients With Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MET-2-201
Record Dates: First submitted 2018-11-21; First posted 2019-02-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2020-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b, placebo-controlled, multiple dose pilot study.
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded as to which dosing arm the subjects are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MET-2 20 g (Experimental): Subjects will be given a once-daily loading dose of 5 grams (g) of MET-2 in the form of 10 MET-2 capsules orally for the first 4 days. For the following 10 days, patients will take 1.5 g MET-2 in the form of three MET-2 capsules taken once-daily
  Interventions: Biological: MET-2
- MET-2 40 g (Experimental): Subjects will be given a once-daily loading dose of 10 g of MET-2 in the form of 20 MET-2 capsules orally for the first 4 days. For the following 10 days, subjects will take 1.5 g MET-2 in the form of three MET-2 capsules taken once daily
  Interventions: Biological: MET-2
- Placebo oral capsule (Placebo Comparator): Subjects receive 10 placebo capsules that are identical in appearance to the MET-2 capsules
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Biological: MET-2 — MET-2 is a defined consortium of human commensal bacteria derived from a healthy donor, which has the full metabolic functional capacity of fecal microbiota.
  Arms: MET-2 20 g; MET-2 40 g
Drug: Placebo oral capsule — Placebo oral capsule which is identical to the MET-2 capsules.
  Arms: Placebo oral capsule

SUMMARY:
To define the parameters for dose-dependent engraftment of MET-2 commensal bacteria for the treatment of mild to moderate ulcerative colitis

DETAILED DESCRIPTION:
This study will deliver MET-2 at two different doses via an oral capsule in patients with active mucosal inflammation and observe its safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and clinical efficacy as compared to placebo. The goal is to define the parameters for dose-dependent engraftment of MET-2 commensal bacteria for the treatment of mild to moderate ulcerative colitis not fully responsive to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to Moderate UC.
2. ≥ 18 years old.
3. Able to provide informed consent, or have a caregiver able to provide consent.
4. Subjects must have a documented diagnosis (radiologic or endoscopic with histology) of UC for >3 months before screening. The following must be available in each subject's source documentation:

   * A biopsy report to confirm the histological diagnosis
   * A report documenting disease duration and medication history prior to study colonoscopy
5. Subjects receiving any treatment(s) forUC are eligible provided they are anticipated to be on a stable dose for the duration of the study period and have been on therapy prior to the randomization visit for the following amount of time:

   Prednisone - 4 weeks; Budesonide - 4 weeks; 5-aminosalicylic acid (5-ASA) containing products - 4 weeks; Thiopurine analogs (azathioprine, 6-mercaptopurine) - 12 weeks; Biologic therapy (infliximab, adalimumab, vedolizumab) - 12 weeks; Tofacitinib - 8 weeks.

   No change in dose is permitted for the following time period prior to the randomization visit:

   Prednisone - 2 weeks; Budesonide - 4 weeks; 5-ASA containing products - 4 weeks; Thiopurine analogs (azathioprine, 6-mercaptopurine) - 6 weeks; Biologic therapy (infliximab, adalimumab, vedolizumab) - 6 weeks; Tofacitinib - 4 weeks.
6. Subjects are males or nonpregnant, nonlactating females who, if sexually active, agree to comply with the contraceptive requirements of the protocol, or females of nonchildbearing potential. Males and females of reproductive potential who are sexually active must agree to use acceptable contraception for the duration of the study.
7. Willing to participate in follow up as part of the study.

Exclusion Criteria:

1. Ulcerative colitis with disease limited to only the distal rectum (<5cm from dentate line).
2. Subjects with indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical/histologic findings suggestive of Crohn's disease will be excluded.
3. Subjects with colonic dysplasia or neoplasia. (Subjects with prior history of adenomatous polyps will be eligible if the polyps have been completely removed).
4. Subjects with toxic megacolon or hospitalized for ulcerative colitis.
5. Subjects with colonic stricture, past medical history of colonic resection, a history of bowel surgery within 6 months before screening, or who are likely to require surgery for UC during the treatment period.
6. Use of antibiotics within 6 weeks of randomization visit.
7. Allergy to vancomycin.
8. Elective surgery that will require preoperative antibiotics planned within 3 months of enrolment.
9. Pregnant or planning to get pregnant in the next 6 months.
10. Any condition for which, in the opinion of the investigator, the subject should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome restoration | Baseline vs. day 42
  Microbiologic assessment of fecal deoxyribonucleic acid (DNA) samples will be obtained before, during and after treatment to quantify the change in microbial alpha diversity using statistical methods such as Shannon Diversity Index and Microbiome Health Index

SECONDARY OUTCOMES:
Assessment of mucosal healing | Baseline vs. Day 42
  Mucosal biopsies will be taken and assessed. Assessment will be made using the Mayo Score for Ulcerative Colitis. There are four domains in this scale: Stool frequency, Rectal bleeding, Findings on endoscopy, Physician's global assessment. Each domain has a scoring range of 0 - 3, where 0 represents best possible outcome and 3 represents worst possible outcome. Efficacy of treatment will be defined as a 'Findings on endoscopy' score of less than or equal to one.
Inflammatory Bowel Disease Questionnaire | Baseline vs. Day 42
  This is a self-administered questionnaire. There are 32 quality of life questions related to bowel function. Each question is rated on a numerical scale. The number of possible ratings varies between questions but is most frequently from 1 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Allan H Steinhart, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided